CLINICAL TRIAL: NCT00139191
Title: A Pilot Study Evaluating the Correlation Between Carbon 11 Acetate (C-11 Acetate) Uptake and Retention as Measured by Positron Emission Tomography (PET) and Fatty Acid Synthase (FAS) Expression in Prostate Cancer
Brief Title: Study Evaluating the Correlation Between C-11 Acetate Uptake and Retention as Measured by PET and FAS in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-136
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; positron emission tomography; carbon 11 acetate; PET; fatty acid synthase; FAS
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: C-11 acetate PET scan

SUMMARY:
The purpose of this study is to understand if a new type of radiology test called positron emission tomography (PET) with carbon 11 acetate will help us to understand which cancers produce more of a protein called fatty acid synthase (FAS).

DETAILED DESCRIPTION:
* Within 4 weeks of the patient's scheduled surgery they will undergo a C11 acetate PET scan. This scan will be performed at the Massachusetts General Hospital's Nuclear Medicine Department and involves an intravenous injection of acetate with a radioactive tracer followed by a PET scan. The scan will determine how well the tumor is taking up the acetate.
* Patients will also undergo a CT scan of the pelvis at the same time as the PET scan.
* After surgery, the removed tumor will have additional testing that will look at different factors that may tell us how aggressive the tumor is and how much FAS is within the tumor. FAS seems to be produced in higher amounts by prostate cancer cells than normal cells. We will then try to determine if the results of the C11 acetate PET scan can tell us how much FAS is produced by prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented prostate cancer
* Planned radical prostatectomy
* > 50% cores positive for prostate cancer from prostate biopsy or a palpable prostate nodule
* Older than 18 years of age

Exclusion Criteria:

* Inability to lay on a scanner for 60 minutes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To explore the associations between measures of C-11 acetate uptake and retention into prostate tumors and levels of FAS expression in tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts